CLINICAL TRIAL: NCT01613976
Title: A Phase Ib, Open-label, Multi-center, Dose-escalation Study of Oral Panobinostat (LBH589) Administered With 5-Azacitidine (Vidaza®) in Adult Japanese Patients With Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMML) or Acute Myeloid Leukemia (AML)
Brief Title: A Phase Ib Study of Panobinostat (LBH589) in Combination With 5-Azacitidine for Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMML) or Acute Myeloid Leukemia (AML) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589H1101
Record Dates: First submitted 2012-05-24; First posted 2012-06-07 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Myelodysplastic Syndromes (MDS); Chronic Myelomonocytic Leukemia (CMML); Acute Myeloid Leukemia (AML)
Keywords: Myelodysplastic Syndromes; MDS; Chronic Myelomonocytic Leukemia; CMML; Acute Myeloid Leukemia; AML; Panobinostat; LBH589; 5-Aza; Azacitidine
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panobinostat and Azacitidine (Experimental): combination regimen
  Interventions: Drug: Panobinostat

INTERVENTIONS:
Drug: Panobinostat
  Other Names: LBH589

SUMMARY:
The purpose of this study is to confirm the safety and tolerability of oral panobinostat (PAN) in combination with a fixed dose of 5-Azacitidine (5-Aza) in adult Japanese patients with Myelodysplastic Syndromes (MDS), Chronic Myelomonocytic Leukemia (CMML) or Acute Myeloid Leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

1. Japanese patients who are candidates for treatment with 5-Aza and present with one of the following:

   * intermediate-2 or high-risk MDS according to the International Prognostic Scoring System (IPSS). OR
   * AML with multilineage dysplasia and maximum of 30% blasts (former RAEB-T according to FAB) OR CMML
2. Patient has an ECOG performance status of ≤ 2
3. Patients must have the following laboratory values unless elevations are considered due to MDS or leukemia: AST/SGOT and/or ALT/SGPT ≤ 2.5 x ULN; serum creatinine ≤ 1.5 x ULN; serum bilirubin (total and direct) ≤ 2 x ULN; electrolyte panel without clinically relevant abnormalities

Exclusion Criteria:

1. Patient who is planned for or has history of hematopoietic stem-cell transplantation (HSCT)
2. Patients with relapsed/refractory AML
3. Patient is receiving concurrent anti-cancer therapy
4. Patient has received prior treatment with deacetylase inhibitors (DACi)
5. Patient has received prior treatment with 5-Aza or 6-aza-2'-deoxycytidine (decitabine)

7. Patient has shown suspected hypersensitivity to 5-Aza or Mannitol 8. Patients with impaired cardiac function 9. Patient taking medications with relative risk of prolonging the QT interval or inducing Torsade de pontes if such treatment cannot be discontinued or switched to a different medication prior to starting study treatment 10. Patients with clinical evidence of relevant mucosal or internal bleeding 11. Patient has any other concurrent severe and/or uncontrolled medical conditions

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicitiy(DLT) | first 5 weeks of treatment period
  DLT will be assessed during PK run-in period (up to 7 days) and 1st cycle (28 days)

SECONDARY OUTCOMES:
PK parameter - Cmax | Day 1 to 3 of PK run-in period; pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 24 and 48 hours
PK parameter - Tmax | Day 1 to 3 of PK run-in period; pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 24 and 48 hours
PK parameter - AUC (AUC0-48, AUC0-tlast) | Day 1 to 3 of PK run-in period; pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 24 and 48 hours
PK parameter - T1/2 (apparent oral clearance, volume distribution) | Day 1 to 3 of PK run-in period; pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 24 and 48 hours
PK parameter - AUC0-inf | Day 1 to 3 of PK run-in period; pre-dose (0 hour), 0.5, 1, 2, 3, 4, 6, 8, 24 and 48 hours
Trough level of PAN in combination with 5-Aza | Day 4, 5, 8 of the 1st cycle; pre-dose (0 hour)
Frequency and severity of Adverse Events (AEs) | Participants will be followed for the duration of treatment, an expected average of 6 months
  Safety will be measured in terms of type, frequency and severity of adverse events according to CTCAE v4.03.
Laboratory abnormalities | duration of treatment, an expected average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Japan (5):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Kyoto

REFERENCES:
- [Derived] Kobayashi Y, Munakata W, Ogura M, Uchida T, Taniwaki M, Kobayashi T, Shimada F, Yonemura M, Matsuoka F, Tajima T, Yakushijin K, Minami H. Phase I study of panobinostat and 5-azacitidine in Japanese patients with myelodysplastic syndrome or chronic myelomonocytic leukemia. Int J Hematol. 2018 Jan;107(1):83-91. doi: 10.1007/s12185-017-2327-9. Epub 2017 Sep 13. PMID 28905323
- See also: Novartis results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13549